CLINICAL TRIAL: NCT02839733
Title: Dopamine and Motor Learning in Cerebral Palsy
Status: Terminated | Type: Observational
Why Stopped: Study closed due to change in personnel.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160149; 16-CC-0149
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: Brain Imaging; Adult; DNA Testing; Children; Natural History
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Palsy: Children and young adults with Cerebral Palsy.
- Healthy Volunteer: Children and young adults healthy volunteer

SUMMARY:
Background:

Cerebral palsy (CP) is the most common childhood motor disability. The neurotransmitter dopamine (DA) is important in cognition and emotions/behavior. DA may also be important in motor skill learning. Genes that relate to DA function may affect a person s ability to learn new cognitive or motor skills. Some children with CP can learn motor skills easily while others have trouble. Researchers want to find out if DA gene variations cause some of this variability.

Objectives:

To learn more about how DA and its related genes affect motor and cognitive learning in people with and without CP.

Eligibility:

People ages 5 25 with and without CP who can:

Follow the protocol

Attend and perform the training sessions

Design:

Participants will be screened with:

Medical history

Physical exam

Blood draw for genetic tests

The study has 2 parts. Participants with CP can join both. Those without can join only Part 1.

All participants will have a baseline assessment: short motor skills test and blood draw.

Part 1:

Two 10-session training programs over 2 weeks. Cognitive training will be 2 sessions at the clinic, 8 at home. Participants will perform memory tasks on a computer. All 10 motor training sessions are at the clinic. Participants will step on lines in a virtual reality environment.

Part 2:

Two lab training sessions at least 1 week apart. Participants will perform tasks on a

computer.

Participants with CP may have a brain MRI at 1 visit. They will lie on a table that slides into a machine that takes pictures. They will be in the scanner about 45 minutes. They may have a

DETAILED DESCRIPTION:
Objective

The broad objective of this study is to determine the relationship between variations in genes related to dopamine (DA) neurotransmission in areas of the brain associated with motor leaning (e.g. DRD1, DRD2, DRD3, COMT, DAT) and/or to activity-dependent brain plasticity (e.g. BDNF) and differences in motor learning rates and cognitive processing abilities in persons with and without cerebral palsy (CP). We hypothesize that individual genetic differences will be related to the ability to learn new motor and cognitive skills and may thus provide a potential explanation for the often reported response variability to rehabilitative therapies seen in CP. We will also explore whether motor and cognitive learning abilities are correlated within individuals which could suggest similar underlying neural mechanisms. Finally we would like to evaluate the effect of rewards on procedural learning in those with and without CP, to preliminarily assess how behavioral manipulations of the DA system may affect learning.

Study Population: A maximum of 120 ambulatory children and young adults with and without CP (ages 5-25 inclusive) will be enrolled in this protocol.

Design: This protocol will consist of two separate but related studies: Study #1 is an observational trial whereby subjects with and without CP will participate in two different training paradigms, 10 sessions each, one that involves learning novel working memory tasks and one that involves motor skill learning in the lower extremities, adapted from the horizontal ladder task utilized in rodent studies. All will have blood draws for genetic analyses at baseline, the results of which will be related to changes in performance (learning) per task after training.

Study #2 will be a within-subjects evaluation in CP and controls on the effects of reward (versus no-reward) during learning, which is presumed to increase dopamine transmission. Mean and individual responses to reward-based learning will be assessed and related to genetic variations in dopamine transmission.

For subjects with CP, we would like to obtain brain MRI but this is optional and if they are unable or unwilling to do this portion, they can still participate in this protocol.

Outcome Measures: Primary outcomes are changes in performance (learning) on each task after training which will be related to presence or absence of polymorphisms that have been associated with brain plasticity or with deficits in working memory and/or motor learning. Individual responses to rewards will also be related to variations related to high versus low dopamine transmission in the brain.

ELIGIBILITY:
* INCLUSION CRITERIA:

For all subjects:

1. Ages 5-25 inclusive
2. Able to follow the study protocol
3. Able to attend or perform the training sessions as scheduled

Additional criteria for subjects with CP:

1. Diagnosis of cerebral palsy
2. Gross Motor Functional Classification Scale Level I-II (able to walk at least 10 meters without an assistive device)

EXCLUSION CRITERIA:

For all subjects:

1. Presence of an injury or other medical condition (besides CP) that would affect motor function or the ability to perform the motor training program.

Additional criteria for subjects with CP:

1. Less than 6 months after major surgery to their legs
2. Currently taking levodopa, trihexyphenidyl, methylphenidate or baclofen since these may affect dopamine transmission or neuroplasticity.

Additional criteria for those with CP who choose to have an MRI:

1. Have any of the following contraindications to having an MRI scan:

1. Pregnancy
2. A ventriculo-peritoneal shunt
3. Have claustrophobia and not comfortable in small enclosed spaces
4. Have metal that would make an MRI scan unsafe such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion devise, cochlear or ear implant, transdermal medication patch (nitroglycerine), any metallic implants or objects, body piercing that cannot be removed, bone or joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal embedded (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near your eyes).
5. Excessive startle reaction to or fear of loud noises

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A maximum of 120 ambulatory children and young adults with and without CP (ages 5-25 inclusive) will be enrolled in this protocol.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Learning (specific measures vary by task) | measure of learning of each training task across the entire training period
  There will be two tasks : 1 a motor task which involves walking across a horizontal ladder. 2. Computer base tasks targeting working memory and procedural learning
Genetic testing (for dopamine and activity-related genes) | genetic analyses of individual variations
  COMT, BDNF, DAT, and DRD1, DRD2, DRD3

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Only data without participants protected health information or identifiers will be shared.

REFERENCES:
- [Background] Qian Y, Chen M, Forssberg H, Diaz Heijtz R. Genetic variation in dopamine-related gene expression influences motor skill learning in mice. Genes Brain Behav. 2013 Aug;12(6):604-14. doi: 10.1111/gbb.12062. Epub 2013 Jul 17. PMID 23819855
- [Background] Pearson-Fuhrhop KM, Minton B, Acevedo D, Shahbaba B, Cramer SC. Genetic variation in the human brain dopamine system influences motor learning and its modulation by L-Dopa. PLoS One. 2013 Apr 17;8(4):e61197. doi: 10.1371/journal.pone.0061197. Print 2013. PMID 23613810
- [Background] Molina-Luna K, Pekanovic A, Rohrich S, Hertler B, Schubring-Giese M, Rioult-Pedotti MS, Luft AR. Dopamine in motor cortex is necessary for skill learning and synaptic plasticity. PLoS One. 2009 Sep 17;4(9):e7082. doi: 10.1371/journal.pone.0007082. PMID 19759902
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0149.html